CLINICAL TRIAL: NCT05568121
Title: A Randomized, Open-label, Single-dose, Two-sequence, Two-period, Cross-over Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of L04TD1 and L04RD1 in Healthy Adult Volunteers
Brief Title: A Bioequivalence Study of L04TD1 Compared to Administration of L04RD1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L04-101
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (L04RD1 -> L04TD1) (Experimental): Administration of 1 tablet of L04RD1, and taking 7-day wash-out period, and then administration of 1 tablet of L04TD1
  Interventions: Drug: L04RD1; Drug: L04TD1
- B (L04TD1 -> L04RD1) (Experimental): Administration of 1 tablet of L04TD1, and taking 7-day wash-out period, and then administration of 1 tablet of L04RD1
  Interventions: Drug: L04TD1; Drug: L04RD1

INTERVENTIONS:
Drug: L04RD1 — 1 tablet of L04RD1
  Arms: A (L04RD1 -> L04TD1)
Drug: L04TD1 — 1 tablet of L04TD1
  Arms: A (L04RD1 -> L04TD1)
Drug: L04TD1 — 1 tablet of L04TD1
  Arms: B (L04TD1 -> L04RD1)
Drug: L04RD1 — 1 tablet of L04RD1
  Arms: B (L04TD1 -> L04RD1)

SUMMARY:
This is a randomized, open, single-dose, crossover-design, phase 1, single-center study to evaluate bioequivalence after administration of L04RD1 or administration of L04TD1 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A subject who weighs 50 kg or more at the screening visit and has a body mass index (BMI) of 18.0~29.9 kg/m2
* A subject who is judged to be eligible to participate by the results of screening tests (vital signs, clinical laboratory tests, 12-lead ECG, etc.) by the principal investigator within 30 days before the first administration of the investigational drug
* A subject and their partner who agree to use a medically appropriate method of contraception to exclude potential of pregnancy and not to provide sperm or ova from the first dose to 28 days after the last dose of the investigational drug
* A subject who voluntarily signs the consent form after hearing and understanding the purpose and content of this study, thge characteristics of the investigational drugs, expected adverse reactions, and etc.

Exclusion Criteria:

* A subject who has a history or present symptoms of clinically significant liver, kidney, nervous system, respiratory system, digestive system, endocrine system, blood/tumor, urinary system, cardiovascular system, musculoskeletal disease, or psychiatric disease
* A subject who has an acute illness within 30 days prior to the first dose of investigational drug
* A subject who has a history of gastrointestinal surgery that may affect drug absorption (except simple appendectomy or hernia surgery) or has gastrointestinal diseases
* A subject who has taken drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month prior to the first administration
* A subject who has participated in other clinical trials or bioequivalence studies within 6 months prior to the first dose of the investigational drug
* A subject who is judged unsuitable to participate in this study by the principal investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
AUCt | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
Cmax | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours

SECONDARY OUTCOMES:
AUCinf (Area under the plasma concentration-time curve from time 0 to infinity) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
Tmax (Time of peak plasma concentration) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
AUCt/AUCinf | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
t1/2 (Half-life) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
CL/F | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, South Korea